CLINICAL TRIAL: NCT06618482
Title: Effects of Kinesiotape or Neuromuscular Taping on the Activation of the Transversus Abdominis Muscle. A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Iria Da Cuña Carrera, PHD, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KINESIO2024
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy Subjects (HS)
Keywords: Kinesiotape; Bandage; Transverse Abdominal; Abdominal Ultrasound

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low back kinesiotaping (Experimental)
  Interventions: Procedure: Kinesiotaping
- Transversus abdominis Kinesiotaping (Experimental)
  Interventions: Procedure: Kinesiotaping

INTERVENTIONS:
Procedure: Kinesiotaping — Low back kinesiotaping
  Other Names: neuromuscular bandage
  Arms: Low back kinesiotaping
Procedure: Kinesiotaping — Transversus abdominis kinesiotaping
  Other Names: neuromuscular bandage
  Arms: Transversus abdominis Kinesiotaping

SUMMARY:
The use of adhesive bandages is a widely practiced technique in both clinical and sports settings. There is a great variety of materials used for bandaging, with multiple objectives: limiting movement, correcting joint positions, reducing pain, enhancing sports performance, and reducing the number of injuries.

However, current knowledge about their potential effects is still limited, and more studies are needed to determine the most appropriate application parameters.

For this reason, the objective of the study for which we request your collaboration is to determine to what extent the application of an adhesive bandage (neuromuscular tape) can influence muscle facilitation through fiber recruitment and strength development, to improve performance during exercise.

The information derived from this research will provide a better understanding of the influence that an adhesive bandage (neuromuscular tape) can have on the neuromuscular system and on strength enhancement.

DETAILED DESCRIPTION:
Kinesiotape (KT) or neuromuscular tape is an adhesive elastic bandage developed in Japan by Kenzo Kase in the 1970s. It became widely known during the 2008 Beijing Olympics when it was used by multiple professional athletes. It is a therapeutic tool used in physiotherapy for the treatment of musculoskeletal injuries and other conditions. The design of this tape aims to mimic the characteristics of the skin in weight, thickness, and flexibility. It is made of 100% cotton, which facilitates evaporation and quick drying, allowing it to be worn for up to 5 days.

Kase et al. proposed several benefits depending on the application method: providing positional stimulus through the skin, aligning fascial tissues, increasing subcutaneous space in an area of inflammation, assisting or limiting movement, and eliminating edema through the lymphatic channels. These benefits are attributed to analgesic effects, proprioceptive effects, increased blood and lymphatic flow, and muscle tone regulation.

There is controversy over the ability of this tape to induce muscle activation or inhibition. A previous study suggests that KT does not have a significant effect on muscle strength, while others advocate its use for muscle facilitation due to observed increases in strength and performance.

On the other hand, interest in spinal stability in the rehabilitation area, understood as the spine's ability to resist disturbances, has increased in recent decades. The "core" or stabilizing muscles include those of the back, abdomen, pelvic floor, diaphragm, hips, and glutes. They are responsible for transferring forces from the proximal to the distal areas of the body, thus considered protective elements in performing functional tasks (most activities require dynamic balance) and generating large torques by the limbs.

Core stability work is mainly applied in sports performance, spinal conditions, and lumbar pain associated with instability, pregnancy, and postpartum; although it could be extended to multiple dysfunctions. Regarding patients with lumbar pain, there is evidence of a high correlation with central muscle dysfunction, finding altered recruitment patterns and especially a delay in the activation of the transverse abdominal muscle during limb movement. During pregnancy, the abdominal wall is in a prolonged state of stretching, often weakening the structure and causing the separation of the rectus abdominis muscles, known as abdominal diastasis.

Despite the widespread use of core training, patients have difficulties initiating the contraction of these muscles and effectively activating the deep stabilizing muscles (transverse abdominal muscle, internal oblique muscle, and lumbar multifidus muscles).

Considering the proposed effects of KT, it is believed that this tape could modify the muscle fiber recruitment pattern through mechanoreceptor stimulation and increased afferent input to the central nervous system (CNS). Although several studies have been conducted on the application of KT on the lower limb to increase strength development, evidence on the use of KT in the activation of abdominal muscles is limited.

Some studies apply lumbar KT to test its effect on core activity, with contradictory results. Other studies use KT to stimulate rectus activity and thus reduce abdominal diastasis, obtaining favorable effects.

Few studies use KT on abdominal muscles to stimulate their activation during exercise. Gürşen et al. applied it to the rectus and oblique abdominals in women with cesarean sections, finding a significant increase in strength. Pourahmadi et al. evaluated the immediate effects on abdominal muscle endurance, with applications on the transverse and internal oblique muscles producing short-term improvements. The KT application described in the study for the transverse abdominal muscle is as follows: transverse placement of an I-cut KT strip (50% tension) between the two anterior superior iliac spines (ASIS).

As previously mentioned, KT is a widely used technique, although scientific evidence on its effectiveness is limited and contradictory. While some research focuses on stimulating superficial abdominal muscles, it has not yet been scientifically proven that KT affects the activation of the transverse muscle.

The main objective of this experimental study is to evaluate the effect of stimulating KT application on the transverse abdominal muscle of healthy subjects to determine its activation using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* The participants are members of the UVIGO who voluntarily participate in the study with an age between 18 and 35 years.
* The participants are healthy subjects (men and women) of legal age.
* All subjects must sign the informed consent prior to the experimentation.

Exclusion Criteria:

* - Suffering from skin disorders, fragile skin or allergy to adhesive bandages.
* Elite athletes.
* Excessive skin hair in the region to apply the bandage.
* Receive a bandage in the abdominal or lumbar region two weeks prior to the experiment.
* History of orthopedic/traumatic alterations in the lumbopelvic region (deformities, arthrodesis, arthropathy, muscle injuries, fracture or tendinopathy), neurological disorders (central or peripheral), systemic disorders, circulatory disorders (edema, heart failure, thrombosis, renal failure), or surgery in the abdominal-lumbar region in the last 6 months.
* Perform abdominal or lumbar strength training 48 hours prior to the study.
* Limitation greater than 50% in the flexion-extension range of motion of the lumbar spine.
* Consumption of alcoholic beverages or medications 24 hours prior to the experimentation.
* Pregnancy or having given birth in less than a year.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness of the transverse abdominis muscle | 30 minutes
  Muscle thickness of the transverse abdominis muscle mesured with ultrasound

IPD SHARING:
Plan to Share IPD: No